CLINICAL TRIAL: NCT04169685
Title: Comparison of Dexmedetomidine and Propofol for Sedation in Adult Patients Undergoing Flexible Bronchoscopy -A Retrospective Review
Brief Title: Dexmedetomidine for Sedation Undergoing Bronchoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Sheng-Hua Wu, MD, Kaohsiung Medical University
Other Study IDs: KMUHIRB-E(I)-20190221
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Safety Issues
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with dexmedetomidine: Drugs provided moderate sedation during procedure including dexmedetomidine
  Interventions: Procedure: bronchoscopy
- without dexmedetomidine: Drugs provided moderate sedation during procedure without dexmedetomidine
  Interventions: Procedure: bronchoscopy

INTERVENTIONS:
Procedure: bronchoscopy — during flexible bronchoscopy

SUMMARY:
Several sedatives or analgesics can be used to achieve appropriate levels of sedation for endoscopic procedures. Dexmedetomide is notable for providing sedation without respiratory depression. We hypothesized dexmedetomide is more suitable for sedation of bronchoscopy than other sedative drugs.

DETAILED DESCRIPTION:
A retrospective chart review was conducted. All patients undergoing flexible bronchoscopy with moderate sedation were enrolled.The primary analysis outcome was safety profile during procedure included incidence of procedure interruption, incidence of snoring and observed apnea, transient hypoxemia and hypotension. The secondary outcome was measured by recovery profile (awake and ambulation time).

ELIGIBILITY:
Inclusion Criteria:

* sedation undergoing flexible bronchoscopy

Exclusion Criteria:

* without sedation undergoing flexible bronchoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing flexible bronchoscopy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
safety profile during procedure | during procedure
  Incidence of procedure interruption, incidence of snoring and observed apnea, transient hypoxemia and hypotension

CONTACTS AND LOCATIONS:
Overall Officials: sheng hua wu, MD, PHD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No